CLINICAL TRIAL: NCT00220337
Title: A Multicenter, Open-label Trial to Assess the Long-term Safety and Efficacy of Lacosamide in Subjects With Painful Diabetic Neuropathy
Brief Title: A Trial to Assess the Long-term Safety and Efficacy of Lacosamide in Subjects With Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Collaborators: SCHWARZ BIOSCIENCES GmbH - Part of UCB Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0830; 2004-000960-28 (EudraCT Number)
Record Dates: First submitted 2005-09-01; First posted 2005-09-22 (Estimated); Results first posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2022-08

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Painful diabetic neuropathy; Lacosamide
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Lacosamide; 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

ARMS (1):
- Lacosamide (LCM) (Experimental): Open label active treatment
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Lacosamide film-coated tablets; two times per day; up to 400 mg/day for 2.75 years
  Other Names: SPM 927

SUMMARY:
The purpose of this study is to determine if lacosamide (SPM 927) is safe if taken for a longer period of time and whether it continues to work well to treat pain.

Subjects will receive lacosamide at a dose that will be individually determined to be the one that provides most pain relief with the least side effects. The maximum dose will be 600mg/day. Subjects may participate in this trial until October 2007. This time may be extended to allow them to participate until lacosamide is commercially available.

If a subject meet the requirements for the study at Visit 1 and after a two weeks phase without trial medication, s/he enters a Titration Phase to determine the personal optimal dose of lacosamide. When this dose is reached s/he will enter the Maintenance Phase and will be asked to return for visits every 4 weeks for the first 24 weeks and every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Painful diabetic neuropathy

Exclusion Criteria:

* no clinically relevant liver enzyme abnormalities and impaired renal function, no cardiac abnormalities, no pregnant or nursing females

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2004-12-21; Primary Completion 2007-10-31 (Actual); Study Completion 2007-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB (+1 844 599 2273)
Locations (1):
- Monheim, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in December 2004 and concluded in October 2007.
Pre-assignment Details: Participant Flow refers to the Safety Set.
Groups:
- Lacosamide: Subjects received lacosamide 100 mg (milligrams)/day (50 mg twice daily), orally which was up titrated in increments of 100 mg up to a maximum optimal dose of 400 mg/day during Titration Phase (Weeks 1 to 4). Subjects entered Maintenance Phase after the optimal dose was achieved and received it for up to a maximum of 140 weeks.
Period: Overall Study
Arm/Group | Lacosamide
Started | 371
Completed | 192
Not Completed | 179
Not completed — Adverse Event | 70
Not completed — Lack of Efficacy | 17
Not completed — Withdrawal by Subject | 68
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 5
Not completed — Other | 12
Not completed — Unsatisfactory compliance | 5

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set which consisted of all subjects who received at least 1 dose of study medication.
Groups:
- Lacosamide: Subjects received lacosamide 100 mg/day (50 mg twice daily), orally which was up titrated in increments of 100 mg up to a maximum optimal dose of 400 mg/day during Titration Phase (Weeks 1 to 4). Subjects entered Maintenance Phase after the optimal dose was achieved and received it for up to a maximum of 140 weeks.
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 262
  >=65 years | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181
  Male | 190

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Adverse Events (AE) Reported Spontaneously by the Subject or Observed by the Investigator
Description: An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment.
Time Frame: From Screening until Safety Follow up Visit (up to 140 weeks)
Population: The Safety Set (SS) was defined as all subjects who signed the informed consent form and took at least 1 dose of trial medication.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
percentage of participants | 80.9

2. Primary Outcome: Percentage of Subjects With Marked Abnormalities in Hematology Parameters After Start of Treatment During the Titration Period
Description: Changes in hematology parameters is reported as incidence of marked abnormalities in - Hematocrit (<=.85x Lower Limit Normal [LLN] or >= 1.15x Upper Limit Normal [ULN] - Hemoglobin (<=.85x LLN or >=1.15x ULN) - White Blood Cell (WBC) Count (<=3.0 or >=16.0 G/l) - Basophils (>=5.0%) - Eosinophils (>=10%) - Monocytes (>=20%) - Platelet Count (<=100 or >=600 G/l)
Time Frame: During the titration period (up to Week 8)
Population: Safety Set included 371 subjects. Only subjects with valid data for hematology parameters are included in the analysis. Here, Number analyzed signifies those subjects who were evaluable for different hematologic parameters.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
percentage of participants
  Hematocrit: number analyzed (Participants) | 362
  Hematocrit | 0.8
  Hemoglobin: number analyzed (Participants) | 367
  Hemoglobin | 0.5
  White Blood Cell: number analyzed (Participants) | 366
  White Blood Cell | 1.4
  Basophils: number analyzed (Participants) | 364
  Basophils | 1.1
  Eosinophils: number analyzed (Participants) | 363
  Eosinophils | 0
  Monocytes: number analyzed (Participants) | 366
  Monocytes | 0
  Platelet Count: number analyzed (Participants) | 361
  Platelet Count | 1.1

3. Primary Outcome: Percentage of Subjects With Marked Abnormalities in Hematology Parameters After Start of Treatment During the Maintenance Period
Description: as for outcome 2
Time Frame: During the maintenance period (up to 136 weeks)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
percentage of participants
  Hematocrit: number analyzed (Participants) | 321
  Hematocrit | 6.2
  Hemoglobin: number analyzed (Participants) | 326
  Hemoglobin | 5.5
  WBC Count: number analyzed (Participants) | 325
  WBC Count | 2.8
  Basophils: number analyzed (Participants) | 324
  Basophils | 2.8
  Eosinophils: number analyzed (Participants) | 322
  Eosinophils | 2.8
  Monocytes: number analyzed (Participants) | 325
  Monocytes | 0.3
  Platelet Count: number analyzed (Participants) | 320
  Platelet Count | 4.4

4. Primary Outcome: Percentage of Subjects With Marked Abnormalities Clinical Chemistry Parameters After Start of Treatment During the Titration Period
Description: Changes in clinical chemistry parameters is reported as incidence of marked abnormalities in - Alanine aminotransferase ([ALT] 3x ULN) - Alanine aminotransferase ([ALT] 5x ULN) - Alanine aminotransferase [(ALT] 10x ULN) - Aspartate aminotransferase ([AST] 3x ULN) - Aspartate aminotransferase ([AST] 5x ULN) - Aspartate aminotransferase ([AST] 10x ULN) - Alkaline Phosphatase (3x ULN) - Gamma-glutamyltransferase ([GGT] 3x ULN) - Total Bilirubin (2x ULN) - Albumin (<26 g/l) - Blood Urea Nitrogen (>=14.28 mmol/l) - Creatinine (>=2.0 mg/dl) - Calcium (<=7.6 or >=11.0 mg/dl) - Chloride (<=90 or >=112 mmol/l) - Phosphorus (<=2.0 or >=6.0 mg/dl) - Potassium (<=3.0 or >=6.0 mmol/l) - Sodium (<127 or >151 mmol/l) - Glucose (<50 or >=200 mg/dl) - Total Cholesterol (>6.5 mmol/l) - Uric Acid (>565.06 umol/l)
Time Frame: During the titration period (up to Week 8)
Population: Safety Set included 371 subjects. Only subjects with valid data for clinical chemistry parameters are included in the analysis. Here, Number analyzed signifies those subjects who were evaluable for different clinical chemistry parameters.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
percentage of participants
  ALT 3xULN: number analyzed (Participants) | 368
  ALT 3xULN | 0.5
  ALT 5xULN: number analyzed (Participants) | 368
  ALT 5xULN | 0
  ALT 10xULN: number analyzed (Participants) | 368
  ALT 10xULN | 0
  AST 3xULN: number analyzed (Participants) | 368
  AST 3xULN | 0
  AST 5xULN: number analyzed (Participants) | 368
  AST 5xULN | 0
  AST 10xULN: number analyzed (Participants) | 368
  AST 10xULN | 0
  Alkaline Phosphatase: number analyzed (Participants) | 368
  Alkaline Phosphatase | 0
  GGT 3xULN: number analyzed (Participants) | 356
  GGT 3xULN | 0.6
  Total Bilirubin: number analyzed (Participants) | 367
  Total Bilirubin | 0.5
  Albumin: number analyzed (Participants) | 368
  Albumin | 0
  Blood Urea Nitrogen: number analyzed (Participants) | 368
  Blood Urea Nitrogen | 0.8
  Creatinine: number analyzed (Participants) | 368
  Creatinine | 0
  Calcium: number analyzed (Participants) | 362
  Calcium | 1.7
  Chloride: number analyzed (Participants) | 363
  Chloride | 0.3
  Phosphorus: number analyzed (Participants) | 366
  Phosphorus | 1.4
  Potassium: number analyzed (Participants) | 364
  Potassium | 0.3
  Sodium: number analyzed (Participants) | 368
  Sodium | 0
  Glucose: number analyzed (Participants) | 212
  Glucose | 40.6
  Total Cholesterol: number analyzed (Participants) | 31
  Total Cholesterol | 3.2
  Uric Acid: number analyzed (Participants) | 361
  Uric Acid | 1.1

5. Primary Outcome: Percentage of Subjects With Marked Abnormalities Clinical Chemistry Parameters After Start of Treatment During the Maintenance Period
Description: as for outcome 4
Time Frame: During the maintenance period (up to 136 weeks)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
percentage of participants
  ALT 3xULN: number analyzed (Participants) | 328
  ALT 3xULN | 0.6
  ALT 5xULN: number analyzed (Participants) | 328
  ALT 5xULN | 0.3
  ALT 10xULN: number analyzed (Participants) | 328
  ALT 10xULN | 0
  AST 3xULN: number analyzed (Participants) | 328
  AST 3xULN | 0
  AST 5xULN: number analyzed (Participants) | 328
  AST 5xULN | 0
  AST 10xULN: number analyzed (Participants) | 328
  AST 10xULN | 0
  Alkaline Phosphatase: number analyzed (Participants) | 328
  Alkaline Phosphatase | 0.3
  GGT 3xULN: number analyzed (Participants) | 319
  GGT 3xULN | 4.7
  Total Bilirubin: number analyzed (Participants) | 327
  Total Bilirubin | 0.3
  Albumin: number analyzed (Participants) | 328
  Albumin | 0.3
  Blood Urea Nitrogen: number analyzed (Participants) | 328
  Blood Urea Nitrogen | 2.1
  Creatinine: number analyzed (Participants) | 328
  Creatinine | 0.6
  Calcium: number analyzed (Participants) | 323
  Calcium | 2.5
  Chloride: number analyzed (Participants) | 323
  Chloride | 3.4
  Phosphorus: number analyzed (Participants) | 326
  Phosphorus | 3.4
  Potassium: number analyzed (Participants) | 325
  Potassium | 2.8
  Sodium: number analyzed (Participants) | 328
  Sodium | 0
  Glucose: number analyzed (Participants) | 193
  Glucose | 66.8
  Total Cholesterol: number analyzed (Participants) | 280
  Total Cholesterol | 0.7
  Uric Acid: number analyzed (Participants) | 323
  Uric Acid | 1.5

6. Primary Outcome: Number of Subjects With Urine pH= 5.0 at Baseline, Categorized by Urine pH at Last Visit
Description: Urinalysis was performed locally at all visits using a urine dipstick test. Categories are as following: pH= 5.0, pH= 6.0, pH= 6.5, pH= 7.0, pH= 7.5, pH= 8.0, pH= 8.5, not done (data not available). Baseline value taken at Visit 2 or at screening for parameters not collected at Visit 2. Last visit is the last post-baseline visit observed under exposure of trial medication, including unscheduled visits.
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with urine pH= 5.0 at baseline are included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 239
Participants
  pH= 5.0 | 194
  pH= 6.0 | 35
  pH= 6.5 | 2
  pH= 7.0 | 3
  pH= 7.5 | 1
  pH= 8.0 | 0
  pH= 8.5 | 0
  not done | 4

7. Primary Outcome: Number of Subjects With Urine pH= 6.0 at Baseline, Categorized by Urine pH at Last Visit
Description: as for outcome 6
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with urine pH= 6.0 at baseline are included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 93
Participants
  pH= 5.0 | 52
  pH= 6.0 | 31
  pH= 6.5 | 4
  pH= 7.0 | 2
  pH= 7.5 | 1
  pH= 8.0 | 1
  pH= 8.5 | 0
  not done | 2

8. Primary Outcome: Number of Subjects With Urine pH= 6.5 at Baseline, Categorized by Urine pH at Last Visit
Description: as for outcome 6
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with urine pH= 6.5 at baseline are included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 24
Participants
  pH= 5.0 | 10
  pH= 6.0 | 7
  pH= 6.5 | 5
  pH= 7.0 | 0
  pH= 7.5 | 0
  pH= 8.0 | 1
  pH= 8.5 | 0
  not done | 1

9. Primary Outcome: Number of Subjects With Urine pH= 7.0 at Baseline, Categorized by Urine pH at Last Visit
Description: as for outcome 6
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with urine pH= 7.0 at baseline are included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 8
Participants
  pH= 5.0 | 4
  pH= 6.0 | 3
  pH= 6.5 | 1
  pH= 7.0 | 0
  pH= 7.5 | 0
  pH= 8.0 | 0
  pH= 8.5 | 0
  not done | 0

10. Primary Outcome: Number of Subjects With Urine pH= 7.5 at Baseline, Categorized by Urine pH at Last Visit
Description: as for outcome 6
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with urine pH= 7.5 at baseline are included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 6
Participants
  pH= 5.0 | 3
  pH= 6.0 | 0
  pH= 6.5 | 3
  pH= 7.0 | 0
  pH= 7.5 | 0
  pH= 8.0 | 0
  pH= 8.5 | 0
  not done | 0

11. Primary Outcome: Number of Subjects With Urine pH= 8.0 at Baseline, Categorized by Urine pH at Last Visit
Description: as for outcome 6
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with urine pH= 8.0 at baseline are included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 1
Participants
  pH= 5.0 | 0
  pH= 6.0 | 0
  pH= 6.5 | 1
  pH= 7.0 | 0
  pH= 7.5 | 0
  pH= 8.0 | 0
  pH= 8.5 | 0
  not done | 0

12. Primary Outcome: Number of Subjects With Urine White Blood Cell Count 'Negative' at Baseline, Categorized by Urine White Blood Cell Count at Last Visit
Description: Urinalysis was performed locally at all visits using a urine dipstick test. Categories are as following: negative, trace, positive +, positive ++, positive +++, not done (data not available). Positive categories (+,++,+++) indicate worsening from Baseline.
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with urine White Blood Cell Count 'Negative' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 344
Participants
  negative | 321
  trace | 7
  positive + | 3
  positive ++ | 5
  positive +++ | 1
  not done | 7

13. Primary Outcome: Number of Subjects With Urine White Blood Cell Count 'Trace' at Baseline, Categorized by Urine White Blood Cell Count at Last Visit
Description: as for outcome 12
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with urine White Blood Cell Count 'Trace' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 15
Participants
  negative | 13
  trace | 1
  positive + | 0
  positive ++ | 0
  positive +++ | 1
  not done | 0

14. Primary Outcome: Number of Subjects With Urine White Blood Cell Count 'Positive +' at Baseline, Categorized by Urine White Blood Cell Count at Last Visit
Description: as for outcome 12
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with urine White Blood Cell Count 'Positive +' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 6
Participants
  negative | 3
  trace | 2
  positive + | 0
  positive ++ | 1
  positive +++ | 0
  not done | 0

15. Primary Outcome: Number of Subjects With Urine White Blood Cell Count 'Positive ++' at Baseline, Categorized by Urine White Blood Cell Count at Last Visit
Description: as for outcome 12
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with urine White Blood Cell Count 'Positive ++' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 6
Participants
  negative | 3
  trace | 0
  positive + | 2
  positive ++ | 1
  positive +++ | 0
  not done | 0

16. Primary Outcome: Number of Subjects With Urine Nitrite Status 'Negative' at Baseline, Categorized by Urine Nitrite Status at Last Visit
Description: Urinalysis was performed locally at all visits using a urine dipstick test. Categories are as following: negative, positive, not done (data not available). Positive category indicate worsening from Baseline.
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Nitrite status 'Negative' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 365
Participants
  negative | 353
  positive | 5
  not done | 7

17. Primary Outcome: Number of Subjects With Urine Nitrite Status 'Positive' at Baseline, Categorized by Urine Nitrite Status at Last Visit
Description: as for outcome 16
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Nitrite status 'Positive' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 6
Participants
  negative | 3
  positive | 3
  not done | 0

18. Primary Outcome: Number of Subjects With Urine Urobilinogen Value 3 µmol/l at Baseline, Categorized by Urine Urobilinogen Value at Last Visit
Description: Categories are as following: 3 µmol/l, 16 µmol/l, 33 µmol/l, 66 µmol/l, not done (data not available).
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Urobilinogen value 3 µmol/l at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 361
Participants
  3 µmol/l | 351
  16 µmol/l | 3
  33 µmol/l | 0
  66 µmol/l | 0
  Not done | 7

19. Primary Outcome: Number of Subjects With Urine Urobilinogen Value 16 µmol/l at Baseline, Categorized by Urine Urobilinogen Value at Last Visit
Description: Categories are as following: 3 µmol/l, 16 µmol/l, 33 µmol/l, 66 µmol/l, not done (data not available).
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Urobilinogen value 16 µmol/l at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 9
Participants
  3 µmol/l | 7
  16 µmol/l | 1
  33 µmol/l | 1
  66 µmol/l | 0
  Not done | 0

20. Primary Outcome: Number of Subjects With Urine Urobilinogen Value 66 µmol/l at Baseline, Categorized by Urine Urobilinogen Value at Last Visit
Description: Categories are as following: 3 µmol/l, 16 µmol/l, 33 µmol/l, 66 µmol/l, not done (data not available).
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Urobilinogen value 66 µmol/l at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 1
Participants
  3 µmol/l | 1
  16 µmol/l | 0
  33 µmol/l | 0
  66 µmol/l | 0
  Not done | 0

21. Primary Outcome: Number of Subjects With Urine Protein Status 'Negative' at Baseline, Categorized by Urine Protein Status at Last Visit
Description: as for outcome 12
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Protein status 'Negative' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 317
Participants
  Negative | 292
  Trace | 13
  Positive + | 3
  Positive ++ | 1
  Positive +++ | 2
  Not done | 6

22. Primary Outcome: Number of Subjects With Urine Protein Status 'Trace' at Baseline, Categorized by Urine Protein Status at Last Visit
Description: Urinalysis was performed locally at all visits using a urine dipstick test. Categories are as following: negative, trace, positive +, positive ++, positive +++, not done (data not available). Positive category (+, ++, +++) indicate worsening from Baseline.
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Protein status 'Trace' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 39
Participants
  Negative | 27
  Trace | 7
  Positive + | 4
  Positive ++ | 0
  Positive +++ | 0
  Not done | 1

23. Primary Outcome: Number of Subjects With Urine Protein Status 'Positive +' at Baseline, Categorized by Urine Protein Status at Last Visit
Description: as for outcome 22
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Protein status 'Positive +' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 7
Participants
  Negative | 3
  Trace | 1
  Positive + | 1
  Positive ++ | 2
  Positive +++ | 0
  Not done | 0

24. Primary Outcome: Number of Subjects With Urine Protein Status 'Positive ++' at Baseline, Categorized by Urine Protein Status at Last Visit
Description: as for outcome 22
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Protein status 'Positive ++' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 6
Participants
  Negative | 2
  Trace | 0
  Positive + | 3
  Positive ++ | 0
  Positive +++ | 1
  Not done | 0

25. Primary Outcome: Number of Subjects With Urine Blood Status 'Negative' at Baseline, Categorized by Urine Blood Status at Last Visit
Description: Urinalysis was performed locally at all visits using a urine dipstick test. Categories are as following: negative, trace (N), trace (H), positive +, positive ++, positive +++, not done (data not available). Positive category (+, ++, +++) indicate worsening from Baseline.
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Blood status 'Negative' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 345
Participants
  Negative | 319
  Trace (N) | 7
  Trace (H) | 1
  Positive + | 3
  Positive ++ | 4
  Positive +++ | 4
  Not done | 7

26. Primary Outcome: Number of Subjects With Urine Blood Status 'Trace (N)' at Baseline, Categorized by Urine Blood Status at Last Visit
Description: as for outcome 25
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Blood status 'Trace (N)' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 17
Participants
  Negative | 14
  Trace (N) | 2
  Trace (H) | 0
  Positive + | 1
  Positive ++ | 0
  Positive +++ | 0
  Not done | 0

27. Primary Outcome: Number of Subjects With Urine Blood Status 'Trace (H)' at Baseline, Categorized by Urine Blood Status at Last Visit
Description: as for outcome 25
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Blood status 'Trace (H)' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 6
Participants
  Negative | 4
  Trace (N) | 2
  Trace (H) | 0
  Positive + | 0
  Positive ++ | 0
  Positive +++ | 0
  Not done | 0

28. Primary Outcome: Number of Subjects With Urine Blood Status 'Positive +' at Baseline, Categorized by Urine Blood Status at Last Visit
Description: as for outcome 25
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Blood status 'Positive +' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 1
Participants
  Negative | 1
  Trace (N) | 0
  Trace (H) | 0
  Positive + | 0
  Positive ++ | 0
  Positive +++ | 0
  Not done | 0

29. Primary Outcome: Number of Subjects With Urine Blood Status 'Positive ++' at Baseline, Categorized by Urine Blood Status at Last Visit
Description: as for outcome 25
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Blood status 'Positive ++' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 2
Participants
  Negative | 1
  Trace (N) | 1
  Trace (H) | 0
  Positive + | 0
  Positive ++ | 0
  Positive +++ | 0
  Not done | 0

30. Primary Outcome: Number of Subjects With Urine Ketone Status 'Negative' at Baseline, Categorized by Urine Ketone Status at Last Visit
Description: Urinalysis was performed locally at all visits using a urine dipstick test. Categories are as following: negative, trace (N), trace, small, moderate, not done (data not available).
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Ketone status 'Negative' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 344
Participants
  Negative | 328
  Trace | 8
  Small | 1
  Moderate | 0
  Not done | 7

31. Primary Outcome: Number of Subjects With Urine Ketone Status 'Trace' at Baseline, Categorized by Urine Ketone Status at Last Visit
Description: as for outcome 30
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Ketone status 'Trace' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 21
Participants
  Negative | 19
  Trace | 0
  Small | 2
  Moderate | 0
  Not Done | 0

32. Primary Outcome: Number of Subjects With Urine Ketone Status 'Small' at Baseline, Categorized by Urine Ketone Status at Last Visit
Description: as for outcome 30
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Ketone status 'Small' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 4
Participants
  Negative | 2
  Trace | 2
  Small | 0
  Moderate | 0
  Not Done | 0

33. Primary Outcome: Number of Subjects With Urine Ketone Status 'Moderate' at Baseline, Categorized by Urine Ketone Status at Last Visit
Description: as for outcome 30
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Ketone status 'Moderate' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 2
Participants
  Negative | 2
  Trace | 0
  Small | 0
  Moderate | 0
  Not Done | 0

34. Primary Outcome: Number of Subjects With Urine Bilirubin Status 'Negative' at Baseline, Categorized by Urine Bilirubin Status at Last Visit
Description: Urinalysis was performed locally at all visits using a urine dipstick test. Categories are as following: negative, positive +, positive ++, not done (data not available). Positive category (+, ++) indicate worsening from Baseline.
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Bilirubin status 'Negative' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 360
Participants
  Negative | 351
  Positive + | 2
  Positive ++ | 0
  Not done | 7

35. Primary Outcome: Number of Subjects With Urine Bilirubin Status 'Positive +' at Baseline, Categorized by Urine Bilirubin Status at Last Visit
Description: as for outcome 34
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Bilirubin status 'Positive +' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 8
Participants
  Negative | 8
  Positive + | 0
  Positive ++ | 0
  Not done | 0

36. Primary Outcome: Number of Subjects With Urine Bilirubin Status 'Positive ++' at Baseline, Categorized by Urine Bilirubin Status at Last Visit
Description: as for outcome 34
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Bilirubin status 'Positive ++' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 3
Participants
  Negative | 3
  Positive + | 0
  Positive ++ | 0
  Not done | 0

37. Primary Outcome: Number of Subjects With Urine Glucose Value 'Negative' at Baseline, Categorized by Urine Glucose Value at Last Visit
Description: Categories are as following: negative, 5.5 mmol/l, 14 mmol/l, 28 mmol/l, 55 mmol/l, >= 111 mmol/l, not done (data not available).
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Glucose value 'Negative' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 266
Participants
  Negative | 194
  5.5 mmol/l | 30
  14 mmol/l | 16
  28 mmol/l | 12
  55 mmol/l | 4
  >=111 mmol | 6
  Not Done | 4

38. Primary Outcome: Number of Subjects With Urine Glucose Value 5.5 mmol/l at Baseline, Categorized by Urine Glucose Value at Last Visit
Description: as for outcome 37
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Glucose value 5.5 mmol/l at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 37
Participants
  Negative | 18
  5.5 mmol/l | 15
  14 mmol/l | 2
  28 mmol/l | 1
  55 mmol/l | 0
  >=111 mmol | 0
  Not Done | 1

39. Primary Outcome: Number of Subjects With Urine Glucose Value 14 mmol/l at Baseline, Categorized by Urine Glucose Value at Last Visit
Description: as for outcome 37
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Glucose value 14 mmol/l at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 18
Participants
  Negative | 6
  5.5 mmol/l | 8
  14 mmol/l | 0
  28 mmol/l | 1
  55 mmol/l | 2
  >=111 mmol | 0
  Not Done | 1

40. Primary Outcome: Number of Subjects With Urine Glucose Value 28 mmol/l at Baseline, Categorized by Urine Glucose Value at Last Visit
Description: as for outcome 37
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Glucose value 28 mmol/l at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 20
Participants
  Negative | 10
  5.5 mmol/l | 3
  14 mmol/l | 3
  28 mmol/l | 3
  55 mmol/l | 0
  >=111 mmol | 1
  Not Done | 0

41. Primary Outcome: Number of Subjects With Urine Glucose Value 55 mmol/l at Baseline, Categorized by Urine Glucose Value at Last Visit
Description: as for outcome 37
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Glucose value 55 mmol/l at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 19
Participants
  Negative | 5
  5.5 mmol/l | 5
  14 mmol/l | 1
  28 mmol/l | 3
  55 mmol/l | 1
  >=111 mmol | 4
  Not Done | 0

42. Primary Outcome: Number of Subjects With Urine Glucose Value >=111 mmol/l at Baseline, Categorized by Urine Glucose Value at Last Visit
Description: as for outcome 37
Time Frame: Baseline, Last Visit (up to 140 weeks)
Population: Only subjects with Urine Glucose value >=111 mmol/l at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 11
Participants
  Negative | 3
  5.5 mmol/l | 2
  14 mmol/l | 0
  28 mmol/l | 2
  55 mmol/l | 2
  >=111 mmol | 1
  Not Done | 1

43. Primary Outcome: Percentage of Subjects With Marked Abnormalities in Vital Signs After Start of Treatment
Description: Changes in vital signs examination findings is reported as percentage of subjects with marked abnormalities in - Systolic Blood Pressure (SBP) >=180 mmHg and increase of >=20 mmHg - Systolic Blood Pressure >=90 mmHg and decrease of >=20 mmHg - Diastolic Blood Pressure (DBP) >=105 mmHg and increase of >=15 mmHg - Diastolic Blood Pressure >=50 mmHg and decrease of >=15 mmHg - Pulse Rate (PR) >=120 beats/min and increase of >=15 beats/min - Pulse Rate >=50 beats/min and decrease of >=15 beats/min
Time Frame: During study period (up to 140 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
percentage of participants
  SBP >=180 and increase of >=20 mmHg | 7.5
  SBP <=90 and decrease of >=20 mmHg | 0.3
  DBP >=105 and increase of >=15 mmHg | 3.5
  DBP <=50 and decrease of >=15 mmHg | 0.8
  PR >=120 and increase of >=15 beats/min | 0.3
  PR <=50 and decrease of >=15 beats/min | 0.8

44. Primary Outcome: Percentage of Subjects With Marked Abnormalities in Physical Examination Findings After Start of Treatment.
Description: Changes in physical examination findings is reported as percentage of subjects with marked abnormalities in following categories: - Ears, Eyes, Nose, Mouth, Throat - Cardiovascular - Peripheral vascular - Pulmonary - Musculoskeletal - Hepato- / Gastrointestinal - Renal / Genitourological - Neurological - Metabolic / Endocrine - Psychiatric - Hematological / Lymphatic Nodes - Dermatological - Other The percentages are based on the number of subjects with examinations done at each visit for each body system.
Time Frame: Last Visit (up to 140 weeks)
Population: 371 subjects were included in the safety set. Here, Number analyzed signifies those subjects who were evaluable for prespecified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
percentage of participants
  Ears, Eyes, Nose, Mouth, Throat: number analyzed (Participants) | 329
  Ears, Eyes, Nose, Mouth, Throat | 12.2
  Cardiovascular: number analyzed (Participants) | 330
  Cardiovascular | 15.2
  Peripheral vascular: number analyzed (Participants) | 330
  Peripheral vascular | 14.2
  Pulmonary: number analyzed (Participants) | 329
  Pulmonary | 2.1
  Musculoskeletal: number analyzed (Participants) | 330
  Musculoskeletal | 13.3
  Hepato- / Gastrointestinal: number analyzed (Participants) | 324
  Hepato- / Gastrointestinal | 5.2
  Renal / Genitourological: number analyzed (Participants) | 317
  Renal / Genitourological | 1.3
  Neurological: number analyzed (Participants) | 323
  Neurological | 49.5
  Metabolic / Endocrine: number analyzed (Participants) | 323
  Metabolic / Endocrine | 19.5
  Psychiatric: number analyzed (Participants) | 329
  Psychiatric | 1.5
  Hematological / Lymphatic Nodes: number analyzed (Participants) | 327
  Hematological / Lymphatic Nodes | 0.6
  Dermatological: number analyzed (Participants) | 329
  Dermatological | 16.7
  Other: number analyzed (Participants) | 15
  Other | 93.3

45. Primary Outcome: Percentage of Subjects With Marked Abnormalities in Neurological Examination Findings After Start of Treatment
Description: Changes in neurological examination findings is reported as percentage of subjects with marked abnormalities in following categories: - General - Cranial Nerves - Reflexes - Muscle Strength and Tone - Coordination and Cerebellar Function - Motor System - Sensation: Upper Extremities - Sensation: Lower Extremities The percentages are based on the number of subjects with examinations done at last visit for each category or parameter.
Time Frame: Last Visit (up to 140 weeks)
Population: as for outcome 44
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
percentage of participants
  General: number analyzed (Participants) | 329
  General | 3.6
  Cranial Nerves: number analyzed (Participants) | 329
  Cranial Nerves | 13.4
  Reflexes: number analyzed (Participants) | 326
  Reflexes | 69.9
  Muscle Strength and Tone: number analyzed (Participants) | 328
  Muscle Strength and Tone | 13.4
  Coordination and Cerebellar Function: number analyzed (Participants) | 328
  Coordination and Cerebellar Function | 7.0
  Motor System: number analyzed (Participants) | 323
  Motor System | 3.7
  Sensation: Upper Extremities: number analyzed (Participants) | 327
  Sensation: Upper Extremities | 21.1
  Sensation: Lower Extremities: number analyzed (Participants) | 328
  Sensation: Lower Extremities | 87.5

46. Primary Outcome: Percentage of Subjects With Abnormal Electrocardiogram (ECG) Findings
Description: Changes in 12-lead ECGs is reported as percentage of subjects with abnormal ECG findings categorized in 'Abnormal, possibly insignificant' and 'Abnormal, possibly significant' based on the alert criterion by the ECG vendor and not on the investigator's assessment.
Time Frame: Last Visit (up to 140 weeks)
Population: Only subjects with a last visit assessment who had a normal assessment at Baseline where Baseline is defined as the last ECG assessment prior to the first dose of trial medication are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 150
percentage of participants
  Abnormal, possibly insignificant | 4.7
  Abnormal, possibly significant | 18.0

47. Primary Outcome: Percentage of Subjects Who Withdrew Due to Adverse Events (AEs)
Description: as for outcome 1
Time Frame: During the study period (up to 140 weeks)
Population: The Safety Set was defined as all subjects who signed the informed consent form and took at least 1 dose of trial medication.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
percentage of participants | 16.4

48. Secondary Outcome: Change in Average Pain Interference With Sleep From the Baseline Week to the 7 Days Prior to Each Visit
Description: Pain interference scores at each visit (sleep and activity respectively) were defined as the average of the respective daily interference scores during the 7 last available days prior to the corresponding visit. An 11-point Likert scale was used to assess the subject's sleep. The subject rated how the pain had interfered with sleep over the past 12 hours, from 0 (no interference) to 10 (complete interference). A negative value indicates improvement in symptoms from Baseline. Subjects rated pain interference over the past 12 hours for 7 days prior to each visit and an average value was calculated for each subject.
Time Frame: Baseline, Visit 2.1, Visit 2.2, Visit 2.4, Visit 2.5, Visit 3, Visit 4, Visit 5, Visit 6, Visit 7, Visit 8, Visit 9.0, Visit 9.1, Visit 9.2, Visit 9.3, Visit 9.4, Visit 9.5, Visit 9.6, Visit 9.7, Visit 9.8, Visit 9.9
Population: 371 subjects were included in the Safety set. Only subjects with available data for Pain Interference with sleep at the respective visit are included in the analysis. Here, Number analyzed signifies those subjects who were evaluable for each visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Visit 2.1: number analyzed (Participants) | 368
  Visit 2.1 | -0.99 (1.614)
  Visit 2.2: number analyzed (Participants) | 230
  Visit 2.2 | -1.35 (1.939)
  Visit 2.3: number analyzed (Participants) | 107
  Visit 2.3 | -1.77 (1.916)
  Visit 2.4: number analyzed (Participants) | 10
  Visit 2.4 | -1.25 (1.218)
  Visit 2.5: number analyzed (Participants) | 3
  Visit 2.5 | -1.38 (1.003)
  Visit 3: number analyzed (Participants) | 331
  Visit 3 | -2.62 (2.166)
  Visit 4: number analyzed (Participants) | 330
  Visit 4 | -3.05 (2.313)
  Visit 5: number analyzed (Participants) | 315
  Visit 5 | -3.29 (2.311)
  Visit 6: number analyzed (Participants) | 308
  Visit 6 | -3.27 (2.269)
  Visit 7: number analyzed (Participants) | 299
  Visit 7 | -3.37 (2.307)
  Visit 8: number analyzed (Participants) | 290
  Visit 8 | -3.45 (2.273)
  Visit 9.0: number analyzed (Participants) | 288
  Visit 9.0 | -3.51 (2.328)
  Visit 9.1: number analyzed (Participants) | 274
  Visit 9.1 | -3.44 (2.256)
  Visit 9.2: number analyzed (Participants) | 254
  Visit 9.2 | -3.45 (2.229)
  Visit 9.3: number analyzed (Participants) | 242
  Visit 9.3 | -3.65 (2.154)
  Visit 9.4: number analyzed (Participants) | 233
  Visit 9.4 | -3.56 (2.130)
  Visit 9.5: number analyzed (Participants) | 220
  Visit 9.5 | -3.60 (2.130)
  Visit 9.6: number analyzed (Participants) | 209
  Visit 9.6 | -3.47 (2.247)
  Visit 9.7: number analyzed (Participants) | 197
  Visit 9.7 | -3.54 (2.185)
  Visit 9.8: number analyzed (Participants) | 181
  Visit 9.8 | -3.62 (2.124)
  Visit 9.9: number analyzed (Participants) | 46
  Visit 9.9 | -3.35 (1.875)

49. Secondary Outcome: Change in Average Pain Interference With General Activity From the Baseline Week to the 7 Days Prior to Each Visit
Description: as for outcome 48
Time Frame: as for outcome 48
Population: 371 subjects were included in the Safety set. Only subjects with available data for Pain Interference with general activity at the respective visit are included in the analysis. Here, Number analyzed signifies those subjects who were who were evaluable for each visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Visit 2.1: number analyzed (Participants) | 366
  Visit 2.1 | -0.99 (1.571)
  Visit 2.2: number analyzed (Participants) | 228
  Visit 2.2 | -1.38 (1.827)
  Visit 2.3: number analyzed (Participants) | 106
  Visit 2.3 | -1.66 (1.962)
  Visit 2.4: number analyzed (Participants) | 10
  Visit 2.4 | -1.21 (1.279)
  Visit 2.5: number analyzed (Participants) | 3
  Visit 2.5 | -1.62 (0.951)
  Visit 3: number analyzed (Participants) | 331
  Visit 3 | -2.56 (2.130)
  Visit 4: number analyzed (Participants) | 330
  Visit 4 | -2.97 (2.273)
  Visit 5: number analyzed (Participants) | 313
  Visit 5 | -3.14 (2.292)
  Visit 6: number analyzed (Participants) | 308
  Visit 6 | -3.17 (2.291)
  Visit 7: number analyzed (Participants) | 297
  Visit 7 | -3.27 (2.321)
  Visit 8: number analyzed (Participants) | 290
  Visit 8 | -3.32 (2.317)
  Visit 9.0: number analyzed (Participants) | 288
  Visit 9.0 | -3.45 (2.307)
  Visit 9.1: number analyzed (Participants) | 270
  Visit 9.1 | -3.52 (2.221)
  Visit 9.2: number analyzed (Participants) | 252
  Visit 9.2 | -3.50 (2.123)
  Visit 9.3: number analyzed (Participants) | 242
  Visit 9.3 | -3.62 (2.177)
  Visit 9.4: number analyzed (Participants) | 232
  Visit 9.4 | -3.60 (2.129)
  Visit 9.5: number analyzed (Participants) | 217
  Visit 9.5 | -3.65 (2.116)
  Visit 9.6: number analyzed (Participants) | 208
  Visit 9.6 | -3.50 (2.263)
  Visit 9.7: number analyzed (Participants) | 196
  Visit 9.7 | -3.53 (2.189)
  Visit 9.8: number analyzed (Participants) | 180
  Visit 9.8 | -3.66 (2.158)
  Visit 9.9: number analyzed (Participants) | 46
  Visit 9.9 | -3.56 (1.703)

50. Secondary Outcome: Change in Current Pain From Visit 2 (Baseline) to Each Subsequent Visit as Measured by a 100 mm Visual Analogue Scale (VAS)
Description: A 100 mm visual analogue scale (VAS) was used to assess the subject's current pain. The subject rated their current pain from 0 (no pain) to 100 (worst possible pain). A negative value indicates improvement in symptoms.
Time Frame: as for outcome 48
Population: 371 subjects were included in the Safety set. Only subjects with available data for current pain measured by a 100 mm visual analogue scale (VAS) at the respective visit are included in the analysis. Here, Number of subjects analyzed signifies those subjects who were evaluable for each visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Visit 2.1: number analyzed (Participants) | 365
  Visit 2.1 | -12.32 (19.671)
  Visit 2.2: number analyzed (Participants) | 225
  Visit 2.2 | -20.79 (23.955)
  Visit 2.3: number analyzed (Participants) | 107
  Visit 2.3 | -27.87 (23.218)
  Visit 2.4: number analyzed (Participants) | 10
  Visit 2.4 | -14.80 (14.148)
  Visit 2.5: number analyzed (Participants) | 3
  Visit 2.5 | -20.33 (14.742)
  Visit 3: number analyzed (Participants) | 328
  Visit 3 | -35.23 (24.986)
  Visit 4: number analyzed (Participants) | 325
  Visit 4 | -37.01 (24.952)
  Visit 5: number analyzed (Participants) | 312
  Visit 5 | -37.91 (24.446)
  Visit 6: number analyzed (Participants) | 302
  Visit 6 | -37.71 (24.269)
  Visit 7: number analyzed (Participants) | 297
  Visit 7 | -40.06 (23.653)
  Visit 8: number analyzed (Participants) | 290
  Visit 8 | -40.25 (23.433)
  Visit 9.0: number analyzed (Participants) | 287
  Visit 9.0 | -40.24 (23.739)
  Visit 9.1: number analyzed (Participants) | 275
  Visit 9.1 | -41.47 (22.797)
  Visit 9.2: number analyzed (Participants) | 261
  Visit 9.2 | -40.08 (24.447)
  Visit 9.3: number analyzed (Participants) | 245
  Visit 9.3 | -41.56 (24.140)
  Visit 9.4: number analyzed (Participants) | 234
  Visit 9.4 | -41.00 (22.533)
  Visit 9.5: number analyzed (Participants) | 224
  Visit 9.5 | -41.45 (23.199)
  Visit 9.6: number analyzed (Participants) | 211
  Visit 9.6 | -40.88 (24.142)
  Visit 9.7: number analyzed (Participants) | 197
  Visit 9.7 | -41.69 (23.089)
  Visit 9.8: number analyzed (Participants) | 181
  Visit 9.8 | -41.83 (23.278)
  Visit 9.9: number analyzed (Participants) | 49
  Visit 9.9 | -43.63 (21.543)

51. Secondary Outcome: Percentage of Patients With Categorized Patient's Global Impression of Change in Pain (PGIC) at Visit 4
Description: The PGIC is a 7-point categorical rating scale in which the subject rates the change in his/her pain since starting trial medication. Categories are as following: much worse, moderately worse, mildly worse, no change, mildly better, moderately better, much better.
Time Frame: Visit 4
Population: Only patients with available data for Patient's Global Impression of Change in Pain (PGIC) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 317
percentage of participants
  Much Worse | 0
  Moderately Worse | 0
  Mildly Worse | 0.9
  No Change | 6.0
  Mildly Better | 27.1
  Moderately Better | 32.5
  Much Better | 33.4

52. Secondary Outcome: Percentage of Patients With Categorized Patient's Global Impression of Change in Pain (PGIC) at Visit 6
Description: as for outcome 51
Time Frame: Visit 6
Population: Only patients with available data for Patient's Global Impression of Change in Pain (PGIC) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 299
percentage of participants
  Much Worse | 0
  Moderately Worse | 0
  Mildly Worse | 2
  No Change | 8.4
  Mildly Better | 23.7
  Moderately Better | 34.8
  Much Better | 31.1

53. Secondary Outcome: Percentage of Patients With Categorized Patient's Global Impression of Change in Pain (PGIC) at Visit 9.0
Description: as for outcome 51
Time Frame: Visit 9.0
Population: Only patients with available data for Patient's Global Impression of Change in Pain (PGIC) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 277
percentage of participants
  Much Worse | 0
  Moderately Worse | 0.7
  Mildly Worse | 1.4
  No Change | 6.1
  Mildly Better | 18.8
  Moderately Better | 35.7
  Much Better | 37.2

54. Secondary Outcome: Percentage of Patients With Categorized Patient's Global Impression of Change in Pain (PGIC) at Visit 9.1
Description: as for outcome 51
Time Frame: Visit 9.1
Population: Only patients with available data for Patient's Global Impression of Change in Pain (PGIC) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 269
percentage of participants
  Much Worse | 0.7
  Moderately Worse | 0.4
  Mildly Worse | 2.6
  No Change | 5.6
  Mildly Better | 18.2
  Moderately Better | 37.2
  Much Better | 35.3

55. Secondary Outcome: Percentage of Patients With Categorized Patient's Global Impression of Change in Pain (PGIC) at Visit 9.2
Description: as for outcome 51
Time Frame: Visit 9.2
Population: Only patients with available data for Patient's Global Impression of Change in Pain (PGIC) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 249
percentage of participants
  Much Worse | 0.4
  Moderately Worse | 0.8
  Mildly Worse | 4.0
  No Change | 4.4
  Mildly Better | 17.3
  Moderately Better | 34.5
  Much Better | 38.6

56. Secondary Outcome: Percentage of Patients With Categorized Patient's Global Impression of Change in Pain (PGIC) at Visit 9.3
Description: as for outcome 51
Time Frame: Visit 9.3
Population: Only patients with available data for Patient's Global Impression of Change in Pain (PGIC) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 237
percentage of participants
  Much Worse | 0
  Moderately Worse | 1.3
  Mildly Worse | 3.0
  No Change | 4.2
  Mildly Better | 20.7
  Moderately Better | 34.6
  Much Better | 36.3

57. Secondary Outcome: Percentage of Patients With Categorized Patient's Global Impression of Change in Pain (PGIC) at Visit 9.4
Description: as for outcome 51
Time Frame: Visit 9.4
Population: Only patients with available data for Patient's Global Impression of Change in Pain (PGIC) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 226
percentage of participants
  Much Worse | 0
  Moderately Worse | 0.9
  Mildly Worse | 4.4
  No Change | 5.8
  Mildly Better | 18.6
  Moderately Better | 35.0
  Much Better | 35.4

58. Secondary Outcome: Percentage of Patients With Categorized Patient's Global Impression of Change in Pain (PGIC) at Visit 9.5
Description: as for outcome 51
Time Frame: Visit 9.5
Population: Only patients with available data for Patient's Global Impression of Change in Pain (PGIC) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 212
percentage of participants
  Much Worse | 0
  Moderately Worse | 1.9
  Mildly Worse | 3.3
  No Change | 6.6
  Mildly Better | 18.4
  Moderately Better | 34.4
  Much Better | 35.4

59. Secondary Outcome: Percentage of Patients With Categorized Patient's Global Impression of Change in Pain (PGIC) at Visit 9.6
Description: as for outcome 51
Time Frame: Visit 9.6
Population: Only patients with available data for Patient's Global Impression of Change in Pain (PGIC) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 202
percentage of participants
  Much Worse | 0
  Moderately Worse | 3.0
  Mildly Worse | 1.5
  No Change | 7.9
  Mildly Better | 19.3
  Moderately Better | 31.2
  Much Better | 37.1

60. Secondary Outcome: Percentage of Patients With Categorized Patient's Global Impression of Change in Pain (PGIC) at Visit 9.7
Description: as for outcome 51
Time Frame: Visit 9.7
Population: Only patients with available data for Patient's Global Impression of Change in Pain (PGIC) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 184
percentage of participants
  Much Worse | 0.5
  Moderately Worse | 2.2
  Mildly Worse | 3.8
  No Change | 6.0
  Mildly Better | 20.1
  Moderately Better | 31.5
  Much Better | 35.9

61. Secondary Outcome: Percentage of Patients With Categorized Patient's Global Impression of Change in Pain (PGIC) at Visit 9.8
Description: as for outcome 51
Time Frame: Visit 9.8
Population: Only patients with available data for Patient's Global Impression of Change in Pain (PGIC) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 49
percentage of participants
  Much Worse | 0
  Moderately Worse | 2.0
  Mildly Worse | 4.1
  No Change | 8.2
  Mildly Better | 10.2
  Moderately Better | 36.7
  Much Better | 38.8

62. Secondary Outcome: Percentage of Patients With Categorized Patient's Global Impression of Change in Pain (PGIC) at Termination Visit
Description: as for outcome 51
Time Frame: Termination Visit (last treatment visit)
Population: Only patients with available data for Patient's Global Impression of Change in Pain (PGIC) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 329
percentage of participants
  Much Worse | 0.9
  Moderately Worse | 2.4
  Mildly Worse | 3.6
  No Change | 13.4
  Mildly Better | 20.4
  Moderately Better | 28.6
  Much Better | 30.7

63. Secondary Outcome: Change in Different Symptoms of Neuropathic Pain From Visit 2 (Baseline) to Visit 4
Description: Subjects were asked to assess different symptoms of neuropathic pain with respect to severity using the Neuropathic Pain Symptoms Inventory (NPSI) at different visits. It comprised of 10 descriptive symptom questions (pain feels like burning, squeezing, pressure electric shocks, stabbing, pins/needles, tingling, provoked or increased by brushing, pressure or contact with something cold), and 2 temporal questions (duration of pain, number of pain attacks). The NPSI scores of the descriptive questions are reported in categories below, which were rated on an 11-point scale from 0 (absence of pain) to 10 (maximum intensity of pain). Higher scores indicate a greater intensity of pain. A negative value indicates improvement in symptoms from Baseline. This assessment was done only in subjects from countries in which a validated version of the NPSI was available.
Time Frame: Baseline, Visit 4
Population: 371 subjects were included in the Safety Set. Only patients with available data for different symptoms of neuropathic pain are included in the analysis. Here, Number Analyzed signifies those subjects who were evaluable at prespecified categories.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Burning: number analyzed (Participants) | 109
  Burning | -3.1 (3.00)
  Squeezing: number analyzed (Participants) | 109
  Squeezing | -1.5 (3.53)
  Pressure: number analyzed (Participants) | 108
  Pressure | -2.6 (3.47)
  Electric shocks: number analyzed (Participants) | 109
  Electric shocks | -2.3 (3.41)
  Stabbing: number analyzed (Participants) | 109
  Stabbing | -2.6 (3.56)
  Brushing: number analyzed (Participants) | 109
  Brushing | -1.0 (2.90)
  Increased by pressure: number analyzed (Participants) | 109
  Increased by pressure | -1.9 (3.49)
  Contact with cold: number analyzed (Participants) | 109
  Contact with cold | -1.4 (2.51)
  Pins and needles: number analyzed (Participants) | 109
  Pins and needles | -2.7 (3.36)
  Tingling: number analyzed (Participants) | 109
  Tingling | -2.3 (3.58)

64. Secondary Outcome: Change in Different Symptoms of Neuropathic Pain From Visit 2 (Baseline) to Visit 6
Description: Subjects were asked to assess different symptoms of neuropathic pain with respect to severity using the NPSI at different visits. It comprised of 10 descriptive symptom questions (pain feels like burning, squeezing, pressure electric shocks, stabbing, pins/needles, tingling, provoked or increased by brushing, pressure or contact with something cold), and 2 temporal questions (duration of pain, number of pain attacks). The NPSI scores of the descriptive questions are reported in categories below, which were rated on an 11-point scale from 0 (absence of pain) to 10 (maximum intensity of pain). Higher scores indicate a greater intensity of pain. A negative value indicates improvement in symptoms from Baseline. This assessment was done only in subjects from countries in which a validated version of the NPSI was available.
Time Frame: Baseline, Visit 6
Population: Only patients with available data for different symptoms of neuropathic pain are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 102
units on a scale
  Burning | -2.9 (3.28)
  Squeezing | -1.7 (3.35)
  Pressure | -2.5 (3.10)
  Electric shocks | -2.5 (3.20)
  Stabbing | -2.6 (3.18)
  Brushing | -1.2 (3.12)
  Increased by pressure | -1.8 (3.36)
  Contact with cold | -1.2 (2.90)
  Pins and needles | -3.3 (2.89)
  Tingling | -2.9 (3.58)

65. Secondary Outcome: Change in Different Symptoms of Neuropathic Pain From Visit 2 (Baseline) to Visit 9.0
Description: as for outcome 64
Time Frame: Baseline, Visit 9.0
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Burning: number analyzed (Participants) | 88
  Burning | -3.0 (2.78)
  Squeezing: number analyzed (Participants) | 88
  Squeezing | -2.2 (3.16)
  Pressure: number analyzed (Participants) | 88
  Pressure | -2.7 (3.00)
  Electric shocks: number analyzed (Participants) | 88
  Electric shocks | -2.9 (3.04)
  Stabbing: number analyzed (Participants) | 88
  Stabbing | -2.9 (3.10)
  Brushing: number analyzed (Participants) | 86
  Brushing | -1.0 (2.99)
  Increased by pressure: number analyzed (Participants) | 87
  Increased by pressure | -2.4 (3.13)
  Contact with cold: number analyzed (Participants) | 87
  Contact with cold | -1.2 (3.23)
  Pins and needles: number analyzed (Participants) | 88
  Pins and needles | -3.2 (3.05)
  Tingling: number analyzed (Participants) | 88
  Tingling | -2.9 (3.20)

66. Secondary Outcome: Change in Different Symptoms of Neuropathic Pain From Visit 2 (Baseline) to Visit 9.1
Description: Subjects were asked to assess different symptoms of neuropathic pain with respect to severity using the NPSI at different visits. It comprised of 10 descriptive symptom questions (pain feels like burning, squeezing, pressure electric shocks, stabbing, pins/needles, tingling, provoked or increased by brushing, pressure or contact with something cold), which were rated on an 11-point scale from 0 (absence of pain) to 10 (maximum intensity of pain), and are reported in categories below and 2 temporal questions (duration of pain, number of pain attacks). This assessment was done only in subjects from countries in which a validated version of the NPSI was available. Total NPSI scale ranged from 0 (no pain) to 100 (maximum pain). Higher scores indicate a greater intensity of pain. A negative value indicates improvement in symptoms from Baseline.
Time Frame: Baseline, Visit 9.1
Population: Only patients with available data for different symptoms of neuropathic pain are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 85
units on a scale
  Burning | -3.1 (3.33)
  Squeezing | -2.1 (3.20)
  Pressure | -2.8 (3.10)
  Electric shocks | -3.1 (3.36)
  Stabbing | -2.9 (3.17)
  Brushing | -1.0 (2.92)
  Increased by pressure | -2.3 (3.00)
  Contact with cold | -1.4 (2.78)
  Pins and needles | -3.1 (3.25)
  Tingling | -2.9 (3.33)

67. Secondary Outcome: Change in Different Symptoms of Neuropathic Pain From Visit 2 (Baseline) to Visit 9.2
Description: as for outcome 64
Time Frame: Baseline, Visit 9.2
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Burning: number analyzed (Participants) | 72
  Burning | -3.2 (3.11)
  Squeezing: number analyzed (Participants) | 72
  Squeezing | -2.4 (3.15)
  Pressure: number analyzed (Participants) | 72
  Pressure | -2.7 (3.37)
  Electric shocks: number analyzed (Participants) | 72
  Electric shocks | -2.8 (3.41)
  Stabbing: number analyzed (Participants) | 71
  Stabbing | -3.0 (3.35)
  Brushing: number analyzed (Participants) | 72
  Brushing | -1.0 (2.88)
  Increased by pressure: number analyzed (Participants) | 72
  Increased by pressure | -2.3 (3.00)
  Contact with cold: number analyzed (Participants) | 72
  Contact with cold | -1.7 (2.56)
  Pins and needles: number analyzed (Participants) | 72
  Pins and needles | -3.2 (3.18)
  Tingling: number analyzed (Participants) | 72
  Tingling | -3.0 (3.19)

68. Secondary Outcome: Change in Different Symptoms of Neuropathic Pain From Visit 2 (Baseline) to Visit 9.3
Description: as for outcome 64
Time Frame: Baseline, Visit 9.3
Population: Only patients with available data for different symptoms of neuropathic pain are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 63
units on a scale
  Burning | -3.1 (3.00)
  Squeezing | -1.9 (2.64)
  Pressure | -2.6 (2.82)
  Electric shocks | -3.0 (3.02)
  Stabbing | -2.8 (3.38)
  Brushing | -0.8 (2.88)
  Increased by pressure | -2.5 (3.13)
  Contact with cold | -1.5 (2.88)
  Pins and needles | -2.9 (3.13)
  Tingling | -3.3 (3.44)

69. Secondary Outcome: Change in Different Symptoms of Neuropathic Pain From Visit 2 (Baseline) to Visit 9.4
Description: as for outcome 64
Time Frame: Baseline, Visit 9.4
Population: Only patients with available data for different symptoms of neuropathic pain are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 62
units on a scale
  Burning | -2.8 (2.97)
  Squeezing | -1.5 (2.74)
  Pressure | -2.3 (3.01)
  Electric shocks | -2.3 (3.61)
  Stabbing | -2.8 (3.50)
  Brushing | -0.9 (2.93)
  Increased by pressure | -2.2 (2.97)
  Contact with cold | -1.4 (2.76)
  Pins and needles | -2.8 (3.3)
  Tingling | -3.1 (3.26)

70. Secondary Outcome: Change in Different Symptoms of Neuropathic Pain From Visit 2 (Baseline) to Visit 9.5
Description: as for outcome 64
Time Frame: Baseline, Visit 9.5
Population: Only patients with available data for different symptoms of neuropathic pain are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 59
units on a scale
  Burning | -3.1 (3.09)
  Squeezing | -2.0 (2.86)
  Pressure | -2.4 (2.92)
  Electric shocks | -2.8 (3.20)
  Stabbing | -2.8 (3.36)
  Brushing | -1.0 (2.65)
  Increased by pressure | -2.3 (3.20)
  Contact with cold | -1.6 (2.91)
  Pins and needles | -3.0 (3.20)
  Tingling | -3.1 (3.64)

71. Secondary Outcome: Change in Different Symptoms of Neuropathic Pain From Visit 2 (Baseline) to Visit 9.6
Description: as for outcome 64
Time Frame: Baseline, Visit 9.6
Population: Only patients with available data for different symptoms of neuropathic pain are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 55
units on a scale
  Burning | -3.0 (3.23)
  Squeezing | -2.0 (3.02)
  Pressure | -2.8 (2.84)
  Electric shocks | -3.1 (3.37)
  Stabbing | -2.8 (3.43)
  Brushing | -0.8 (2.55)
  Increased by pressure | -2.7 (3.04)
  Contact with cold | -1.4 (2.65)
  Pins and needles | -3.1 (3.25)
  Tingling | -3.5 (3.31)

72. Secondary Outcome: Change in Different Symptoms of Neuropathic Pain From Visit 2 (Baseline) to Visit 9.7
Description: as for outcome 64
Time Frame: Baseline, Visit 9.7
Population: Only patients with available data for different symptoms of neuropathic pain are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 53
units on a scale
  Burning | -3.2 (3.34)
  Squeezing | -2.1 (3.29)
  Pressure | -2.2 (3.31)
  Electric shocks | -2.9 (3.27)
  Stabbing | -2.5 (3.52)
  Brushing | -1.0 (2.87)
  Increased by pressure | -2.5 (3.12)
  Contact with cold | -1.2 (2.79)
  Pins and needles | -3.2 (3.00)
  Tingling | -3.3 (3.17)

73. Secondary Outcome: Change in Different Symptoms of Neuropathic Pain From Visit 2 (Baseline) to Visit 9.8
Description: as for outcome 64
Time Frame: Baseline, Visit 9.8
Population: Only patients with available data for different symptoms of neuropathic pain are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 19
units on a scale
  Burning | -2.3 (3.43)
  Squeezing | -2.0 (2.89)
  Pressure | -1.7 (2.00)
  Electric shocks | -3.0 (2.65)
  Stabbing | -2.5 (2.82)
  Brushing | -0.4 (2.45)
  Increased by pressure | -1.6 (2.06)
  Contact with cold | -1.4 (1.92)
  Pins and needles | -3.0 (2.94)
  Tingling | -3.2 (3.15)

74. Secondary Outcome: Change in Different Symptoms of Neuropathic Pain From Visit 2 (Baseline) to Termination Visit
Description: as for outcome 64
Time Frame: Baseline, Termination Visit (last treatment visit)
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Burning: number analyzed (Participants) | 116
  Burning | -2.6 (3.47)
  Squeezing: number analyzed (Participants) | 115
  Squeezing | -1.5 (3.20)
  Pressure: number analyzed (Participants) | 115
  Pressure | -2.0 (3.21)
  Electric shocks: number analyzed (Participants) | 116
  Electric shocks | -2.1 (3.54)
  Stabbing: number analyzed (Participants) | 116
  Stabbing | -2.3 (3.45)
  Brushing: number analyzed (Participants) | 116
  Brushing | -1.0 (3.35)
  Increased by pressure: number analyzed (Participants) | 116
  Increased by pressure | -1.8 (3.16)
  Contact with cold: number analyzed (Participants) | 116
  Contact with cold | -0.7 (3.15)
  Pins and needles: number analyzed (Participants) | 116
  Pins and needles | -2.7 (3.36)
  Tingling: number analyzed (Participants) | 116
  Tingling | -2.5 (3.83)

75. Secondary Outcome: Percentage of Subjects With Presence of Spontaneous Pain Categorized by Duration of Pain at Visit 2 (Baseline)
Description: Presence of spontaneous pain was analyzed using the Neuropathic Pain Symptom Inventory (NPSI). This questionnaire comprises 10 descriptive questions, which are rated on 0 to 10 point scales, and 2 temporal questions. Categories of duration of pain are as following: permanently, between 8 and 12 h, between 4 and 7 h, between 1 and 3 h, Less than 1 h. This assessment was done only in subjects from countries in which a validated version of the NPSI was available.
Time Frame: Visit 2 (Baseline)
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 141
percentage of participants
  Permanently | 37.6
  Between 8 and 12 h | 21.3
  Between 4 and 7 h | 19.1
  Between 1 and 3 h | 14.2
  Less than 1 h | 7.8

76. Secondary Outcome: Percentage of Subjects With Presence of Spontaneous Pain Categorized by Duration of Pain at Visit 4
Description: as for outcome 75
Time Frame: Visit 4
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 110
percentage of participants
  Permanently | 10.9
  Between 8 and 12 h | 13.6
  Between 4 and 7 h | 17.3
  Between 1 and 3 h | 20.9
  Less than 1 h | 37.3

77. Secondary Outcome: Percentage of Subjects With Presence of Spontaneous Pain Categorized by Duration of Pain at Visit 6
Description: as for outcome 75
Time Frame: Visit 6
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 103
percentage of participants
  Permanently | 12.6
  Between 8 and 12 h | 7.8
  Between 4 and 7 h | 11.7
  Between 1 and 3 h | 24.3
  Less than 1 h | 43.7

78. Secondary Outcome: Percentage of Subjects With Presence of Spontaneous Pain Categorized by Duration of Pain at Visit 9.0
Description: as for outcome 75
Time Frame: Visit 9.0
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 90
percentage of participants
  Permanently | 11.1
  Between 8 and 12 h | 8.9
  Between 4 and 7 h | 10.0
  Between 1 and 3 h | 22.2
  Less than 1 h | 47.8

79. Secondary Outcome: Percentage of Subjects With Presence of Spontaneous Pain Categorized by Duration of Pain at Visit 9.1
Description: as for outcome 75
Time Frame: Visit 9.1
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 86
percentage of participants
  Permanently | 9.3
  Between 8 and 12 h | 8.1
  Between 4 and 7 h | 15.1
  Between 1 and 3 h | 26.7
  Less than 1 h | 39.5
  Not done | 1.2

80. Secondary Outcome: Percentage of Subjects With Presence of Spontaneous Pain Categorized by Duration of Pain at Visit 9.2
Description: as for outcome 75
Time Frame: Visit 9.2
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 72
percentage of participants
  Permanently | 5.6
  Between 8 and 12 h | 9.7
  Between 4 and 7 h | 8.3
  Between 1 and 3 h | 22.2
  Less than 1 h | 54.2

81. Secondary Outcome: Percentage of Subjects With Presence of Spontaneous Pain Categorized by Duration of Pain at Visit 9.3
Description: as for outcome 75
Time Frame: Visit 9.3
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 64
percentage of participants
  Permanently | 3.1
  Between 8 and 12 h | 3.1
  Between 4 and 7 h | 15.6
  Between 1 and 3 h | 28.1
  Less than 1 h | 50.0

82. Secondary Outcome: Percentage of Subjects With Presence of Spontaneous Pain Categorized by Duration of Pain at Visit 9.4
Description: as for outcome 75
Time Frame: Visit 9.4
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 63
percentage of participants
  Permanently | 6.3
  Between 8 and 12 h | 11.1
  Between 4 and 7 h | 15.9
  Between 1 and 3 h | 22.2
  Less than 1 h | 44.4

83. Secondary Outcome: Percentage of Subjects With Presence of Spontaneous Pain Categorized by Duration of Pain at Visit 9.5
Description: as for outcome 75
Time Frame: Visit 9.5
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 60
percentage of participants
  Permanently | 8.3
  Between 8 and 12 h | 6.7
  Between 4 and 7 h | 15.0
  Between 1 and 3 h | 21.7
  Less than 1 h | 48.3

84. Secondary Outcome: Percentage of Subjects With Presence of Spontaneous Pain Categorized by Duration of Pain at Visit 9.6
Description: as for outcome 75
Time Frame: Visit 9.6
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 56
percentage of participants
  Permanently | 3.6
  Between 8 and 12 h | 10.7
  Between 4 and 7 h | 23.2
  Between 1 and 3 h | 17.9
  Less than 1 h | 44.6

85. Secondary Outcome: Percentage of Subjects With Presence of Spontaneous Pain Categorized by Duration of Pain at Visit 9.7
Description: as for outcome 75
Time Frame: Visit 9.7
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 54
percentage of participants
  Permanently | 7.4
  Between 8 and 12 h | 7.4
  Between 4 and 7 h | 14.8
  Between 1 and 3 h | 16.7
  Less than 1 h | 53.7

86. Secondary Outcome: Percentage of Subjects With Presence of Spontaneous Pain Categorized by Duration of Pain at Visit 9.8
Description: as for outcome 75
Time Frame: Visit 9.8
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 19
percentage of participants
  Permanently | 0
  Between 8 and 12 h | 10.5
  Between 4 and 7 h | 26.3
  Between 1 and 3 h | 26.3
  Less than 1 h | 36.8

87. Secondary Outcome: Percentage of Subjects With Presence of Spontaneous Pain Categorized by Duration of Pain at Termination Visit
Description: as for outcome 75
Time Frame: Termination Visit (last treatment visit)
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 118
percentage of participants
  Permanently | 16.1
  Between 8 and 12 h | 13.6
  Between 4 and 7 h | 16.9
  Between 1 and 3 h | 18.6
  Less than 1 h | 34.7

88. Secondary Outcome: Percentage of Subjects With Pain Attacks in Last the 24 Hours Categorized by Number of Pain Attacks at Visit 2 (Baseline)
Description: Pain attacks were analyzed using the Neuropathic Pain Symptom Inventory (NPSI). This questionnaire comprises 10 descriptive questions, which are rated on 0 to 10 point scales, and 2 temporal questions. Categories of number of pain attacks are as following: no pain attack, between 1 and 5, between 6 and 10, between 11 and 20, more than 20, not done (data not available). This assessment was done only in subjects from countries in which a validated version of the NPSI was available.
Time Frame: Visit 2 (Baseline)
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 141
percentage of participants
  No pain attack | 6.4
  Between 1 and 5 | 33.3
  Between 6 and 10 | 20.6
  Between 11 and 20 | 20.6
  More than 20 | 19.1
  Not done | 0

89. Secondary Outcome: Percentage of Subjects With Pain Attacks in Last the 24 Hours Categorized by Number of Pain Attacks at Visit 4
Description: as for outcome 88
Time Frame: Visit 4
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 110
percentage of participants
  No pain attack | 29.1
  Between 1 and 5 | 39.1
  Between 6 and 10 | 20.9
  Between 11 and 20 | 5.5
  More than 20 | 5.5
  Not done | 0

90. Secondary Outcome: Percentage of Subjects With Pain Attacks in Last the 24 Hours Categorized by Number of Pain Attacks at Visit 6
Description: as for outcome 88
Time Frame: Visit 6
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 104
percentage of participants
  No pain attack | 26.9
  Between 1 and 5 | 42.3
  Between 6 and 10 | 20.2
  Between 11 and 20 | 7.7
  More than 20 | 2.9
  Not done | 0

91. Secondary Outcome: Percentage of Subjects With Pain Attacks in Last the 24 Hours Categorized by Number of Pain Attacks at Visit 9.0
Description: as for outcome 88
Time Frame: Visit 9.0
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 90
percentage of participants
  No pain attack | 36.7
  Between 1 and 5 | 35.6
  Between 6 and 10 | 20.0
  Between 11 and 20 | 5.6
  More than 20 | 2.2
  Not done | 0

92. Secondary Outcome: Percentage of Subjects With Pain Attacks in Last the 24 Hours Categorized by Number of Pain Attacks at Visit 9.1
Description: as for outcome 88
Time Frame: Visit 9.1
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 87
percentage of participants
  No pain attack | 28.7
  Between 1 and 5 | 34.5
  Between 6 and 10 | 20.7
  Between 11 and 20 | 4.6
  More than 20 | 10.3
  Not done | 1.1

93. Secondary Outcome: Percentage of Subjects With Pain Attacks in Last the 24 Hours Categorized by Number of Pain Attacks at Visit 9.2
Description: as for outcome 88
Time Frame: Visit 9.2
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 73
percentage of participants
  No pain attack | 27.4
  Between 1 and 5 | 49.3
  Between 6 and 10 | 9.6
  Between 11 and 20 | 9.6
  More than 20 | 4.1
  Not done | 0

94. Secondary Outcome: Percentage of Subjects With Pain Attacks in Last the 24 Hours Categorized by Number of Pain Attacks at Visit 9.3
Description: as for outcome 88
Time Frame: Visit 9.3
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 63
percentage of participants
  No pain attack | 27.0
  Between 1 and 5 | 44.4
  Between 6 and 10 | 20.6
  Between 11 and 20 | 3.2
  More than 20 | 4.8
  Not done | 0

95. Secondary Outcome: Percentage of Subjects With Pain Attacks in Last the 24 Hours Categorized by Number of Pain Attacks at Visit 9.4
Description: as for outcome 88
Time Frame: Visit 9.4
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 63
percentage of participants
  No pain attack | 31.7
  Between 1 and 5 | 33.3
  Between 6 and 10 | 19.0
  Between 11 and 20 | 11.1
  More than 20 | 4.8
  Not done | 0

96. Secondary Outcome: Percentage of Subjects With Pain Attacks in Last the 24 Hours Categorized by Number of Pain Attacks at Visit 9.5
Description: as for outcome 88
Time Frame: Visit 9.5
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 60
percentage of participants
  No pain attack | 35.0
  Between 1 and 5 | 35.0
  Between 6 and 10 | 21.7
  Between 11 and 20 | 3.3
  More than 20 | 5.0
  Not done | 0

97. Secondary Outcome: Percentage of Subjects With Pain Attacks in Last the 24 Hours Categorized by Number of Pain Attacks at Visit 9.6
Description: as for outcome 88
Time Frame: Visit 9.6
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 56
percentage of participants
  No pain attack | 30.4
  Between 1 and 5 | 44.6
  Between 6 and 10 | 14.3
  Between 11 and 20 | 5.4
  More than 20 | 5.4
  Not done | 0

98. Secondary Outcome: Percentage of Subjects With Pain Attacks in Last the 24 Hours Categorized by Number of Pain Attacks at Visit 9.7
Description: as for outcome 88
Time Frame: Visit 9.7
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 54
percentage of participants
  No pain attack | 33.3
  Between 1 and 5 | 37.0
  Between 6 and 10 | 16.7
  Between 11 and 20 | 5.6
  More than 20 | 7.4
  Not done | 0

99. Secondary Outcome: Percentage of Subjects With Pain Attacks in Last the 24 Hours Categorized by Number of Pain Attacks at Visit 9.8
Description: as for outcome 88
Time Frame: Visit 9.8
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 19
percentage of participants
  No pain attack | 26.3
  Between 1 and 5 | 52.6
  Between 6 and 10 | 15.8
  Between 11 and 20 | 0
  More than 20 | 5.3
  Not done | 0

100. Secondary Outcome: Percentage of Subjects With Pain Attacks in Last the 24 Hours Categorized by Number of Pain Attacks at Termination Visit
Description: as for outcome 88
Time Frame: Termination Visit (last treatment visit)
Population: Only patients with available data for Neuropathic Pain Symptom Inventory (NPSI) are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 118
percentage of participants
  No pain attack | 28.8
  Between 1 and 5 | 35.6
  Between 6 and 10 | 15.3
  Between 11 and 20 | 11.0
  More than 20 | 9.3
  Not done | 0

101. Secondary Outcome: Change in Quality of Life From Visit 2 (Baseline) to Visit 4
Description: Quality of life was analyzed using the Short Form-36 (SF-36) Health Survey quality of life questionnaire. The SF-36 is a participant self-rated questionnaire which consists of 8 sub-scores ranging from 0-100 with higher scores indicating a better health state. The sub-scores are: 1. Physical Functioning, 2. Role-Physical, 3. Bodily Pain, 4. General Health, 5. Vitality, 6. Social Functioning, 7. Role-Emotional, 8. Mental Health. Items 1-4 primarily contribute to the physical component Summary (PCS) score of the SF-36. Items 5-8 primarily contribute to the mental component summary (MCS) score of the SF-36. The PCS and MCS were based on the standardized values of the 8 domains. The maximum and minimum possible values for PCS and MCS is 0-100, where higher scores indicate good condition. A positive value indicates improvement from baseline in quality of life.
Time Frame: Baseline, Visit 4
Population: 371 subjects were included in the Safety Set. Only patients with available data for different sub-scores of SF-36 are included in the analysis. Here, Number Analyzed signifies those subjects who were evaluable at prespecified categories.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Physical Functioning: number analyzed (Participants) | 314
  Physical Functioning | 7.4 (19.99)
  Role-Physical: number analyzed (Participants) | 314
  Role-Physical | 13.1 (39.88)
  Bodily Pain: number analyzed (Participants) | 315
  Bodily Pain | 20.8 (20.14)
  General health: number analyzed (Participants) | 314
  General health | 6.1 (16.18)
  Vitality: number analyzed (Participants) | 315
  Vitality | 8.5 (18.69)
  Social Functioning: number analyzed (Participants) | 315
  Social Functioning | 8.2 (23.79)
  Role-Emotional: number analyzed (Participants) | 314
  Role-Emotional | 7.1 (45.48)
  Mental Health: number analyzed (Participants) | 315
  Mental Health | 5.6 (18.20)
  PCS: number analyzed (Participants) | 312
  PCS | 5.3 (7.62)
  MCS: number analyzed (Participants) | 312
  MCS | 2.2 (10.68)

102. Secondary Outcome: Change in Quality of Life From Visit 2 (Baseline) to Visit 6
Description: Quality of life was analyzed using the SF-36 Health Survey quality of life questionnaire. The SF-36 is a participant self-rated questionnaire which consists of 8 sub-scores ranging from 0-100 with higher scores indicating a better health state. The sub-scores are: 1. Physical Functioning, 2. Role-Physical, 3. Bodily Pain, 4. General Health, 5. Vitality, 6. Social Functioning, 7. Role-Emotional, 8. Mental Health. Items 1-4 primarily contribute to the PCS score of the SF-36. Items 5-8 primarily contribute to the MCS score of the SF-36. The PCS and MCS were based on the standardized values of the 8 domains. The maximum and minimum possible values for PCS and MCS is 0-100, where higher scores indicate good condition. A positive value indicates improvement from baseline in quality of life.
Time Frame: Baseline, Visit 6
Population: as for outcome 101
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Physical Functioning: number analyzed (Participants) | 299
  Physical Functioning | 8.0 (20.55)
  Role-Physical: number analyzed (Participants) | 298
  Role-Physical | 12.1 (39.37)
  Bodily Pain: number analyzed (Participants) | 299
  Bodily Pain | 22.4 (21.02)
  General health: number analyzed (Participants) | 299
  General health | 7.2 (17.48)
  Vitality: number analyzed (Participants) | 299
  Vitality | 8.4 (17.80)
  Social Functioning: number analyzed (Participants) | 299
  Social Functioning | 8.4 (24.47)
  Role-Emotional: number analyzed (Participants) | 299
  Role-Emotional | 8.2 (45.11)
  Mental Health: number analyzed (Participants) | 299
  Mental Health | 5.0 (17.79)
  PCS: number analyzed (Participants) | 298
  PCS | 5.7 (8.13)
  MCS: number analyzed (Participants) | 298
  MCS | 2.2 (10.66)

103. Secondary Outcome: Change in Quality of Life From Visit 2 (Baseline) to Visit 9.0
Description: as for outcome 102
Time Frame: Baseline, Visit 9.0
Population: as for outcome 101
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Physical Functioning: number analyzed (Participants) | 281
  Physical Functioning | 10.4 (21.86)
  Role-Physical: number analyzed (Participants) | 280
  Role-Physical | 17.5 (41.17)
  Bodily Pain: number analyzed (Participants) | 281
  Bodily Pain | 25.3 (20.54)
  General health: number analyzed (Participants) | 279
  General health | 8.8 (16.56)
  Vitality: number analyzed (Participants) | 281
  Vitality | 10.5 (18.89)
  Social Functioning: number analyzed (Participants) | 281
  Social Functioning | 10.3 (25.41)
  Role-Emotional: number analyzed (Participants) | 280
  Role-Emotional | 12.1 (49.96)
  Mental Health: number analyzed (Participants) | 281
  Mental Health | 5.0 (18.01)
  PCS: number analyzed (Participants) | 278
  PCS | 7.1 (7.90)
  MCS: number analyzed (Participants) | 278
  MCS | 2.6 (11.39)

104. Secondary Outcome: Change in Quality of Life From Visit 2 (Baseline) to Visit 9.1
Description: as for outcome 102
Time Frame: Baseline, Visit 9.1
Population: as for outcome 101
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Physical Functioning: number analyzed (Participants) | 268
  Physical Functioning | 10.6 (20.97)
  Role-Physical: number analyzed (Participants) | 267
  Role-Physical | 18.4 (39.92)
  Bodily Pain: number analyzed (Participants) | 268
  Bodily Pain | 24.6 (20.45)
  General health: number analyzed (Participants) | 268
  General health | 7.3 (17.95)
  Vitality: number analyzed (Participants) | 268
  Vitality | 9.6 (18.66)
  Social Functioning: number analyzed (Participants) | 268
  Social Functioning | 10.6 (23.58)
  Role-Emotional: number analyzed (Participants) | 267
  Role-Emotional | 14.7 (47.66)
  Mental Health: number analyzed (Participants) | 268
  Mental Health | 5.6 (17.83)
  PCS: number analyzed (Participants) | 267
  PCS | 6.7 (8.18)
  MCS: number analyzed (Participants) | 267
  MCS | 3.0 (10.83)

105. Secondary Outcome: Change in Quality of Life From Visit 2 (Baseline) to Visit 9.2
Description: as for outcome 102
Time Frame: Baseline, Visit 9.2
Population: as for outcome 101
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Physical Functioning: number analyzed (Participants) | 247
  Physical Functioning | 9.6 (21.54)
  Role-Physical: number analyzed (Participants) | 247
  Role-Physical | 19.2 (42.94)
  Bodily Pain: number analyzed (Participants) | 248
  Bodily Pain | 23.8 (21.33)
  General health: number analyzed (Participants) | 247
  General health | 6.7 (18.83)
  Vitality: number analyzed (Participants) | 248
  Vitality | 9.7 (19.08)
  Social Functioning: number analyzed (Participants) | 248
  Social Functioning | 9.9 (24.79)
  Role-Emotional: number analyzed (Participants) | 247
  Role-Emotional | 13.9 (48.28)
  Mental Health: number analyzed (Participants) | 248
  Mental Health | 6.7 (18.18)
  PCS: number analyzed (Participants) | 245
  PCS | 6.3 (8.31)
  MCS: number analyzed (Participants) | 245
  MCS | 3.3 (11.39)

106. Secondary Outcome: Change in Quality of Life From Visit 2 (Baseline) to Visit 9.3
Description: as for outcome 102
Time Frame: Baseline, Visit 9.3
Population: as for outcome 101
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Physical Functioning: number analyzed (Participants) | 238
  Physical Functioning | 10.3 (21.03)
  Role-Physical: number analyzed (Participants) | 237
  Role-Physical | 20.2 (42.35)
  Bodily Pain: number analyzed (Participants) | 238
  Bodily Pain | 26.3 (21.60)
  General health: number analyzed (Participants) | 238
  General health | 8.3 (17.29)
  Vitality: number analyzed (Participants) | 238
  Vitality | 9.9 (18.40)
  Social Functioning: number analyzed (Participants) | 238
  Social Functioning | 9.8 (24.74)
  Role-Emotional: number analyzed (Participants) | 237
  Role-Emotional | 14.8 (50.82)
  Mental Health: number analyzed (Participants) | 238
  Mental Health | 5.1 (18.52)
  PCS: number analyzed (Participants) | 237
  PCS | 7.2 (8.03)
  MCS: number analyzed (Participants) | 237
  MCS | 2.7 (11.76)

107. Secondary Outcome: Change in Quality of Life From Visit 2 (Baseline) to Visit 9.4
Description: as for outcome 102
Time Frame: Baseline, Visit 9.4
Population: as for outcome 101
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Physical Functioning: number analyzed (Participants) | 225
  Physical Functioning | 9.3 (21.35)
  Role-Physical: number analyzed (Participants) | 224
  Role-Physical | 17.3 (45.59)
  Bodily Pain: number analyzed (Participants) | 225
  Bodily Pain | 24.1 (22.76)
  General health: number analyzed (Participants) | 224
  General health | 6.8 (18.43)
  Vitality: number analyzed (Participants) | 225
  Vitality | 8.7 (19.70)
  Social Functioning: number analyzed (Participants) | 225
  Social Functioning | 9.0 (28.04)
  Role-Emotional: number analyzed (Participants) | 224
  Role-Emotional | 12.1 (49.30)
  Mental Health: number analyzed (Participants) | 225
  Mental Health | 5.0 (18.17)
  PCS: number analyzed (Participants) | 223
  PCS | 6.4 (8.63)
  MCS: number analyzed (Participants) | 223
  MCS | 2.4 (11.74)

108. Secondary Outcome: Change in Quality of Life From Visit 2 (Baseline) to Visit 9.5
Description: as for outcome 102
Time Frame: Baseline, Visit 9.5
Population: as for outcome 101
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
percentage of participants
  Physical Functioning: number analyzed (Participants) | 213
  Physical Functioning | 8.6 (20.88)
  Role-Physical: number analyzed (Participants) | 212
  Role-Physical | 19.1 (45.41)
  Bodily Pain: number analyzed (Participants) | 213
  Bodily Pain | 25.9 (22.49)
  General health: number analyzed (Participants) | 211
  General health | 7.9 (18.64)
  Vitality: number analyzed (Participants) | 213
  Vitality | 7.5 (18.55)
  Social Functioning: number analyzed (Participants) | 213
  Social Functioning | 8.2 (25.00)
  Role-Emotional: number analyzed (Participants) | 212
  Role-Emotional | 9.9 (51.74)
  Mental Health: number analyzed (Participants) | 213
  Mental Health | 3.7 (17.51)
  PCS: number analyzed (Participants) | 210
  PCS | 7.0 (8.53)
  MCS: number analyzed (Participants) | 210
  MCS | 1.4 (11.29)

109. Secondary Outcome: Change in Quality of Life From Visit 2 (Baseline) to Visit 9.6
Description: as for outcome 102
Time Frame: Baseline, Visit 9.6
Population: as for outcome 101
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Physical Functioning: number analyzed (Participants) | 203
  Physical Functioning | 8.6 (21.46)
  Role-Physical: number analyzed (Participants) | 202
  Role-Physical | 18.4 (46.02)
  Bodily Pain: number analyzed (Participants) | 203
  Bodily Pain | 24.8 (22.45)
  General health: number analyzed (Participants) | 203
  General health | 7.0 (18.18)
  Vitality: number analyzed (Participants) | 203
  Vitality | 7.9 (18.39)
  Social Functioning: number analyzed (Participants) | 203
  Social Functioning | 8.8 (24.60)
  Role-Emotional: number analyzed (Participants) | 202
  Role-Emotional | 12.7 (48.39)
  Mental Health: number analyzed (Participants) | 203
  Mental Health | 4.9 (18.78)
  PCS: number analyzed (Participants) | 202
  PCS | 6.5 (8.79)
  MCS: number analyzed (Participants) | 202
  MCS | 2.3 (11.51)

110. Secondary Outcome: Change in Quality of Life From Visit 2 (Baseline) to Visit 9.7
Description: as for outcome 102
Time Frame: Baseline, Visit 9.7
Population: as for outcome 101
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Physical Functioning: number analyzed (Participants) | 184
  Physical Functioning | 9.4 (21.60)
  Role-Physical: number analyzed (Participants) | 183
  Role-Physical | 18.6 (46.18)
  Bodily Pain: number analyzed (Participants) | 184
  Bodily Pain | 25.3 (22.4)
  General Health: number analyzed (Participants) | 184
  General Health | 7.1 (19.13)
  Vitality: number analyzed (Participants) | 184
  Vitality | 7.4 (19.87)
  Social Functioning: number analyzed (Participants) | 184
  Social Functioning | 8.7 (26.12)
  Role-Emotional: number analyzed (Participants) | 183
  Role-Emotional | 8.2 (54.47)
  Mental Health: number analyzed (Participants) | 184
  Mental Health | 4.3 (17.44)
  PCS: number analyzed (Participants) | 183
  PCS | 7.0 (8.62)
  MCS: number analyzed (Participants) | 183
  MCS | 1.4 (11.93)

111. Secondary Outcome: Change in Quality of Life From Visit 2 (Baseline) to Visit 9.8
Description: as for outcome 102
Time Frame: Baseline, Visit 9.8
Population: as for outcome 101
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Physical Functioning: number analyzed (Participants) | 49
  Physical Functioning | 6.9 (23.22)
  Role-Physical: number analyzed (Participants) | 49
  Role-Physical | 2.0 (41.09)
  Bodily Pain: number analyzed (Participants) | 49
  Bodily Pain | 22.2 (20.13)
  General health: number analyzed (Participants) | 49
  General health | 0.2 (20.85)
  Vitality: number analyzed (Participants) | 49
  Vitality | 3.2 (22.95)
  Social Functioning: number analyzed (Participants) | 49
  Social Functioning | 4.3 (26.21)
  Role-Emotional: number analyzed (Participants) | 49
  Role-Emotional | -7.5 (52.38)
  Mental Health: number analyzed (Participants) | 49
  Mental Health | 3.3 (19.48)
  PCS: number analyzed (Participants) | 49
  PCS | 4.6 (8.33)
  MCS: number analyzed (Participants) | 49
  MCS | -0.9 (12.92)

112. Secondary Outcome: Change in Quality of Life From Visit 2 (Baseline) to Termination Visit
Description: as for outcome 102
Time Frame: Baseline, Termination Visit (last treatment visit)
Population: as for outcome 101
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 371
units on a scale
  Physical Functioning: number analyzed (Participants) | 323
  Physical Functioning | 5.0 (22.90)
  Role-Physical: number analyzed (Participants) | 322
  Role-Physical | 7.8 (41.56)
  Bodily Pain: number analyzed (Participants) | 322
  Bodily Pain | 19.3 (23.63)
  General Health: number analyzed (Participants) | 320
  General Health | 4.1 (18.72)
  Vitality: number analyzed (Participants) | 319
  Vitality | 4.5 (18.96)
  Social Functioning: number analyzed (Participants) | 322
  Social Functioning | 4.2 (25.94)
  Role-Emotional: number analyzed (Participants) | 320
  Role-Emotional | 2.5 (51.05)
  Mental Health: number analyzed (Participants) | 319
  Mental Health | 1.2 (18.72)
  PCS: number analyzed (Participants) | 317
  PCS | 4.7 (8.44)
  MCS: number analyzed (Participants) | 317
  MCS | 0.1 (11.41)

113. Primary Outcome: Number of Subjects With Urine Protein Status 'Positive +++' at Baseline, Categorized by Urine Protein Status at Last Visit
Description: as for outcome 22
Time Frame: Last Visit (up to 140 weeks)
Population: Only subjects with Urine Protein status 'Positive +++' at baseline are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 2
Participants
  Negative | 0
  Trace | 0
  Positive + | 0
  Positive ++ | 1
  Positive +++ | 1
  Not done | 0

ADVERSE EVENTS:
Time Frame: From Baseline through Safety follow up visit (up to 140 weeks)
Arm/Group | Lacosamide
All-Cause Mortality (participants affected / at risk) | 7/371
Serious Adverse Events (participants affected / at risk) | 83/371
Other Adverse Events (participants affected / at risk) | 229/371
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lacosamide (N=371)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1
Myocardial infarction (Cardiac disorders) | 3
Angina pectoris (Cardiac disorders) | 2
Myocardial ischaemia (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Pericardial haemorrhage (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Bundle branch block right (Cardiac disorders) | 1
Bundle branch block left (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Vestibular disorder (Ear and labyrinth disorders) | 2
Primary hyperaldosteronism (Endocrine disorders) | 1
Retinal detachment (Eye disorders) | 2
Diabetic retinopathy (Eye disorders) | 2
Cataract (Eye disorders) | 2
Vitreous haemorrhage (Eye disorders) | 1
Eye haemorrhage (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Cataract diabetic (Eye disorders) | 1
Corneal degeneration (Eye disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 2
Pancreatitis acute (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Multi-organ failure (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Biliary colic (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Prostatic abscess (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Diabetic gangrene (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Pubic rami fracture (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Brain herniation (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Investigation (Investigations) | 1
Echocardiogram abnormal (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Diabetic foot (Metabolism and nutrition disorders) | 2
Diabetes mellitus non-insulin- dependent (Metabolism and nutrition disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Toe deformity (Musculoskeletal and connective tissue disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 3
Carotid artery stenosis (Nervous system disorders) | 2
Neuritis (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Syncope vasovagal (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Lumbosacral plexus lesion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Stent placement (Surgical and medical procedures) | 1
Gastric banding (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 3
Circulatory collapse (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Femoral arterial stenosis (Vascular disorders) | 1
Arterial haemorrhage (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lacosamide (N=371)
Nasopharyngitis (Infections and infestations) | 43
Influenza (Infections and infestations) | 21
Back pain (Musculoskeletal and connective tissue disorders) | 26
Dizziness (Nervous system disorders) | 75
Headache (Nervous system disorders) | 44
Somnolence (Nervous system disorders) | 34
Tremor (Nervous system disorders) | 24
Hypertension (Vascular disorders) | 26
Vertigo (Ear and labyrinth disorders) | 45
Nausea (Gastrointestinal disorders) | 49
Vomiting (Gastrointestinal disorders) | 21
Fatigue (General disorders) | 31
Oedema peripheral (General disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days